CLINICAL TRIAL: NCT04100564
Title: Prehospital Airway Control Trial : A Randomized Controlled Trial of Prehospital Airway Management Strategy for Trauma Patients
Brief Title: LITES Task Order 0005 Prehospital Airway Control Trial (PACT)
Acronym: PACT
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Jason Sperry (Other)
Collaborators: United States Department of Defense (U.S. Federal Agency)
Responsible Party: Sponsor-Investigator, Jason Sperry, Professor, University of Pittsburgh
Organization: University of Pittsburgh (Other)
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: STUDY20110369; W81XWH- 16-D- 0024 (Other Grant/Funding Number: Department of Defense)
Record Dates: First submitted 2019-09-11; First posted 2019-09-24 (Actual); Last update posted 2025-11-20 (Actual); Status verified 2025-11

CONDITIONS: Trauma Injury; Airway Control
Keywords: intubation; supraglottic airway
MeSH Terms: conditions — Accidental Injuries

STUDY DESIGN:
Intervention Model Description: Stepped-wedge
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- Standard airway method arm (Active Comparator): Standard airway management strategy
  Interventions: Other: Standard airway management
- Supraglottic airway method arm (Experimental): Supraglottic first airway management strategy
  Interventions: Device: Supraglottic airway device

INTERVENTIONS:
Device: Supraglottic airway device — Initial advanced airway management with a supraglottic device
  Other Names: LMA; King; igel
  Arms: Supraglottic airway method arm
Other: Standard airway management — Initial advanced airway management with standard care method
  Arms: Standard airway method arm

SUMMARY:
The Prehospital Airway Control Trial (PACT) is a proposed 5 year, open label, multi-center, stepped-wedge randomized trial comparing airway management strategies of prehospital trauma patients. The initial airway attempt will be randomized to either usual care (control) or a supraglottic airway management approach (intervention). The primary outcome will be 24 hour survival, with secondary outcomes to include survival to hospital discharge, expected clinical adverse events, airway management performance, ICU length of stay, ventilator days, incidence of ARDS, and incidence of ventilator associated pneumonia. Subjects will be enrolled across approximately 17 prehospital agencies at select LITES Network sites and will enroll a total of 2,009 subjects.

ELIGIBILITY:
Inclusion Criteria:

1. Traumatic injury requiring advanced airway management. Indicators of need for advanced airway management include: a) GCS<8, b) SpO2<90 despite supplemental oxygen, b) ETCO2>60 despite supplemental ventilation, or d) provider discretion.
2. Transport (or intended transport) to an enrolling LITES Trauma Center

Exclusion Criteria:

1. < 15 years of age
2. Known pregnancy
3. Known prisoner
4. Initial advanced airway attempted by a non-PACT provider.
5. Cardiac Arrest without return of spontaneous circulation (ROSC) at the time of the intervention
6. Caustic substance ingestion
7. Airway burns
8. Objection to study voiced by subject or family member at the scene.

Inclusion and exclusion criteria will be assessed based on information available at the time of enrollment, defined as the time at which enrolling agency provides positive pressure ventilation support. Although all reasonable efforts will be made by the emergency medical crew to either directly witness or obtain documentation of inclusion criteria, due to the nature of the emergency prehospital setting, there may be occasions where the emergency medical crew must rely on verbal report of inclusion criteria from referring hospital or emergency crew. In these instances, if, after subsequent review of outside hospital and/or ground crew documentation, it is determined that the subject did not meet inclusion criteria and/or met exclusion criteria, the subject will remain enrolled in the study based on the intention-to-treat principle.

If a verbal report must be used in lieu of physical documentation or directly witnessing inclusion criteria, documentation of the verbal report will serve as the source documentation for determining eligibility. Verbal reports will be documented in the emergency medical record and will detail the information provided and by whom.

Min Age: 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 2009 (Estimated)
Dates: Start 2021-04-01 (Actual); Primary Completion 2026-02 (Estimated); Study Completion 2027-01 (Estimated)

PRIMARY OUTCOMES:
24-hour survival | From injury through 24 hours

SECONDARY OUTCOMES:
Proportion of subjects that survive to hospital discharge | From hospital admission through death or hospital discharge up to 30 days
Rate of first pass success of placement of advanced airway device | At time of placement of device through confirmation of device placement
ICU length of stay | Admission through 30 days or discharge
Ventilator days | Admission through 30 days or discharge
Incidence of expected adverse events | From initial airway management through first 24 hours of hospital admission
Incidence of need for rescue airway device | At the time of placement of device through time of arrival to trauma bay
Incidence of hypoxia | At the time of placement of device through time of arrival to trauma bay
Incidence of hypotension | At the time of placement of device through time of arrival to trauma bay

CONTACTS AND LOCATIONS:
Overall Officials: Jason Sperry, MD, MPH, Principal Investigator — University of Pittsburgh; Francis Guyette, MD, MPH, Principal Investigator — University of Pittsburgh
Locations (14):
- United States (14):
  - Emory University, Atlanta, Georgia
  - Mount Sinai Hospital, Chicago, Illinois
  - Northwestern Memorial Hospital, Chicago, Illinois
  - John H. Stroger Hospital of Cook County, Chicago, Illinois
  - University of Chicago, Chicago, Illinois
  - University of Louisville, Louisville, Kentucky
  - Tulane University, New Orleans, Louisiana
  - Washington University at St. Louis, St Louis, Missouri
  - East Carolina University, Greenville, North Carolina
  - Oregon Health & Science University, Portland, Oregon
  - Allegheny General Hospital, Pittsburgh, Pennsylvania
  - University of Pittsburgh, Pittsburgh, Pennsylvania
  - UPMC, Pittsburgh, Pennsylvania
  - Vanderbilt University, Nashville, Tennessee

IPD SHARING:
Plan to Share IPD: No